CLINICAL TRIAL: NCT04496869
Title: Psychological Impact of COVID19 Among Women Undergoing Infertility Treatment, a French Cohort
Brief Title: Psychological Impact of COVID19 Among Women Undergoing Infertility Treatment
Acronym: PsyCovART
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL20_0577
Record Dates: First submitted 2020-06-15; First posted 2020-08-03 (Actual); Last update posted 2021-07-13 (Actual); Status verified 2021-05

CONDITIONS: Infertility Treatment; Women
Keywords: psychological response; infertility treatment; lockdown period

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Online questionnaire — the investigators sent by email a Googleform online questionnaires to women followed in ART center of HFME (Hospital Femme-Mère-Enfant) . Questions are about demographic characteristics, ART history, feeling during the lockdown. To evaluate psychological impact, the investigators use PSS10 and HADS scales. Both scales are worldwide validated and used in recent COVID19's research. the investigators add some quantitative questions about de feeling during the look down, ART interruption, pregnancy desire.

SUMMARY:
In France, one couple in eight encounters difficulties to conceive. The diagnosis of infertility frequently leads to symptoms of anxiety and depression. These symptoms appear to be higher than in the general population.

Some recent studies have looked at the relationship between anxiety and depression in ART cares.

Results are controversial, but it appears that patients with lower levels of anxiety and depression have higher pregnancy rates. Moreover, in couple, women seem to have more symptoms of anxiety and depression than men.

First epidemiological studies related to the COVID 19 pandemic have shown strong psychological impact on the general population with an anxiety rate estimated at more than 30%.

With COVID 19 pandemic and cessation of ART, it is highly likely that psychic symptoms of anxiety or even depression may have appeared or worsened in women undergoing infertility treatment.

ELIGIBILITY:
Inclusion Criteria:

* Consulting the center between 01/01/2020 to 12/31/2020
* Email address in the medical records
* All causes of infertility

Exclusion Criteria:

* Women followed for:
* Preservation of fertility
* Oocyte donation
* Women who do not speak or read French

Ages: 18 Years to 43 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Women between 18 and 42 years and 12 months, followed in the infertility Center of Femme Mère Enfant Hospital (HFME - Bron - France).
Sampling Method: Non-Probability Sample
Enrollment: 435 (Actual)
Dates: Start 2020-07-07 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2020-08-31 (Actual)

PRIMARY OUTCOMES:
Psychological impact assessed by scores of PSS10 scales. | baseline
  Perceived Stress Scale 10 assess stress in 10 questions with score from 0 to 40. The higher the score is, the more important the stress level is.
Psychological impact assessed by scores of HADS scales. | baseline
  depression Scale with 14 questions. It assesses separately anxiety (score from 0 to 21) and depression (score from 0 to 21).The higher the score is, the more important the anxiety level is.

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Femme Mère Enfant, Bron, France